CLINICAL TRIAL: NCT06117384
Title: Systems Oncology Approach to Optimize Ovarian Cancer Treatment
Acronym: ONCOSYS-OVA
Status: Recruiting | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anniina Färkkilä, Assistant Professor, Specialist in Gynecology, University of Helsinki
Other Study IDs: HUS33342021
Record Dates: First submitted 2023-10-21; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Biomolecular profiling — Molecular and functional analysis of biospecimens, including tumor-normal Whole-exome sequencing, bulk and single-cell RNAsequencing, spatial proteomics, functional testing.

SUMMARY:
The overall aim is to identify effective therapeutic strategies to ovarian cancer (OC) using serial tumor, ascites and blood samples, and carry out state-of-the-art sequencing approaches, functional assays and associated bioinformatics to understand mechanisms behind chemoresistance in OC and identify new treatment options for OC patients. In this observational trial, we will systematically collect, analyze and interpret functional, molecular and clinical data from real-world ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ovarian cancer
* Available tumor tissue/blood samples

Exclusion Criteria:

* Inability to consent to the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All ovarian cancer patients who give their informed consent to the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment and collection of real-world clinical data from ovarian cancer patients | 5 years
  Prospective recruitment and collection of clinical data from 500 ovarian cancer patients. Fraction of patients from which the collection of clinical data including patient age, tumor stage, histological diagnoses have been collected.
Successful collection and translational analysis of biospecimens | 5 years
  Fraction of the recruited patients, from which tumor, ascites, and/or peripheral blood samples that have been successfully collected and subjected to molecular profiling.

SECONDARY OUTCOMES:
Discovery of candidate prognostic and predictive biomarkers | 5 years
  Number of clinical and/or molecular features which of statistically significantly correlate to patient treatment outcomes (response to chemotherapy by RECIST1.1, Progression Free survival, Overall Survival).

CONTACTS AND LOCATIONS:
Overall Officials: Anniina Färkkilä, MD PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University and Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No